CLINICAL TRIAL: NCT03206424
Title: Pattern of Complementary Feeding and Its Impact on Growth Parameters of Infants Under the Age of 2 Years in Assiut Governorate
Brief Title: Patterns of Complementary Feeding in Infancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed maher, Principal Investigator, Assiut University
Other Study IDs: Complementary feeding
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Complementary Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WHO and UNICEF recommend exclusive breastfeeding for six months and addition of complementary foods (CF) at six months of age with continued breastfeeding till two years But WHO estimates that 2 out of 5 children are stunted in low-income countries, so CF should be timely, adequate and prepared and given in a safe manner.

DETAILED DESCRIPTION:
World Health Organization (WHO) and United Nations Children's Fund (UNICEF) recommend exclusive breastfeeding (EBF) for six months, i.e. 180 days and addition of complementary foods at six months of age with continued breastfeeding till at least two years.

When breast milk is no longer enough to meet the nutritional needs of the infant, complementary foods should be added to the diet of the child. The transition from exclusive breastfeeding to family foods, referred to as complementary feeding, typically covers the period from 6 to 18-24 months of age, and is a very vulnerable period.

It is the time when malnutrition starts in many infants, contributing significantly to the high prevalence of malnutrition in children less than five years of age world-wide. WHO estimates that 2 out of 5 children are stunted in low-income countries.

Complementary feeding should be timely, meaning that all infants should start receiving foods in addition to breast milk from 6 months onwards.

It should be adequate, meaning that the complementary foods should be given in amounts, frequency and consistency and using a variety of foods to cover the nutritional needs of the growing child while maintaining breastfeeding.

Foods should be prepared and given in a safe manner, meaning that measures are taken to minimize the risk of contamination with pathogens. And they should be given in a way that is appropriate, meaning that foods are of appropriate texture for the age of the child and applying responsive feeding following the principles of psycho-social care.

Breastfeeding is common in developing countries, but exclusive breastfeeding is rare, and complementary foods are introduced at an early age. Poorer nutritional status was significantly associated with earlier complementary feeding. The results suggest that exclusive breastfeeding, (together with promotion of weaning education and growth monitoring) should be vigorously promoted in these developing countries.

Child development experts advise parents not to introduce solid foods, such as baby cereal, into an infant's diet until the infant is at least 4 to 6 months old. The researchers also found that formula-fed infants were much more likely to be given solid foods too early than were breast-fed infants. Health authorities do advise parents to wait until after 4 months because infants aren't developmentally ready to eat solid foods before. There are a number of other reasons why experts don't recommend early feeding. One is that the early introduction of solid foods has been linked to a shorter duration of breast-feeding. Early solid food consumption has also been linked to the development of chronic conditions, such as childhood obesity, celiac disease, diabetes and eczema.

So that we will do this study in our government region to evaluate Complementary feeding practices and their impact on the health status of our infants, we will recruit a cross sectional sample from those who visit our hospital clinics for various reasons such routine check-ups, vaccinations or illness.

ELIGIBILITY:
Inclusion Criteria:

1. Infants (Age < 2 years).
2. Full Term and Appropriate for Gestational Age (AGA).
3. Infants with successful breastfeeding.

Exclusion Criteria:

1-Children (Age> 2 years). 2. Preterm infants, Small for Gestational Age (SGA) or Intrauterine Growth Retardation (IUGR).

3. Infants with chronic illness, intrauterine infection and major congenital anomalies.

Max Age: 2 Years | Sex: All
Age Groups: Child
Study Population: collecting data through face-to-face interviews with mothers in the health centers for good history and assessment of the infant growth and development.The index cases visiting our hospital and other local public health centers for various reasons such routine check-ups, vaccinations or illness are recruited in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
A questionnaire developed following the guidelines of WHO for CF practices, is used for collecting data through face-to-face interviews with mothers in the health centers. | 16 months
  Specific values taken by good history from mother of the index infant including:
  1. When and why did the mother start complementary feeding?
  2. What is the type of food?
  3. How much food taken in one meal and How many meals are taken within the day?
  4. How does she prepare and give this food?
  5. What the effect of this food on breastfeeding demand or frequency?
  6. Ask about incidence and frequency of problems related to beginning of complementary food such as attacks of Acute gastroenteritis, Constipation or Acute chest infection.
  7. Information about the index infant: name, age, sex, his/her order in the family, height and weight of child at birth.
  8. General information about the parents such as name, age, place of residence, educational level, occupational status, socioeconomic level, self-hygiene and number of children of the family.
  Data will be processed and analyzed using ( Statistical Package for the Social Sciences ) software, version 17
Growth parameters | 16 months
  1. Weight for age percentile.
  2. Height / Length for age percentile.
  3. Weight for Height percentile.
  4. Head Circumference for age percentile.
  Data will be processed and analyzed using ( Statistical Package for the Social Sciences ) software, version 17
Motor development parameters | 16 months
  Motor development milestones will be measured according to the infant actual age:
  1. Head support.
  2. Sitting.
  3. Standing.
  4. Walking.
  5. Running.
  Data will be processed and analyzed using ( Statistical Package for the Social Sciences ) software, version 17
Mental development parameters | 16 months
  Mental development milestones will be measured according to the infant actual age:
  1. Follows moving objects and light.
  2. Laughs loudly and prefers social content.
  3. Recognizes and prefers mother.
  4. Says "Mama, Dada".
  5. Speaks first real word.
  6. Speaks 10-15 words.
  7. Speaks 2- 3 word sentences.
  Data will be processed and analyzed using ( Statistical Package for the Social Sciences ) software, version 17

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Abdellatif, professor, Study Chair — Assuit University- pediatric hospital; Osama M Al-asheer, professor, Study Director — Assuit University - pediatric hospital; Ahmed M Abdullah, resident, Principal Investigator — Assuit University - pediatric hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saleh F, Ara F, Hoque MA, Alam MS. Complementary feeding practices among mothers in selected slums of Dhaka city: a descriptive study. J Health Popul Nutr. 2014 Mar;32(1):89-96. PMID 24847597
- [Result] Batal M, Boulghourjian C, Akik C. Complementary feeding patterns in a developing country: a cross-sectional study across Lebanon. East Mediterr Health J. 2010 Feb;16(2):180-6. PMID 20799572
- [Result] WHO Multicentre Growth Reference Study Group. Complementary feeding in the WHO Multicentre Growth Reference Study. Acta Paediatr Suppl. 2006 Apr;450:27-37. doi: 10.1111/j.1651-2227.2006.tb02373.x. PMID 16817676
- [Result] Davies-Adetugbo AA, Adetugbo K. Effect of early complementary feeding on nutritional status in term infants in rural Nigeria. Nutr Health. 1997;12(1):25-31. doi: 10.1177/026010609701200103. PMID 9403879
- See also: Complementary feeding practices among mothers in selected slums of Dhaka city: a descriptive study — https://www.ncbi.nlm.nih.gov/pubmed/24847597
- See also: Complementary feeding patterns in developing country: a cross-sectional study across Lebanon — https://www.ncbi.nlm.nih.gov/pubmed/?term=Complementary+feeding+patterns+in+developing+country%3A+a+cross-sectional+study+across+Lebanon)+(+Eastern+Mediterranean+Health+Journal).
- See also: WHO Multicentre Growth Reference Study Group. Complementary feeding in the WHO Multicentre Growth Reference Study — https://www.ncbi.nlm.nih.gov/pubmed/16817676
- See also: . Effect of early complementary feeding on nutritional status in term infants in rural Nigeria. Nutr Health — https://www.ncbi.nlm.nih.gov/pubmed/?term=Effect+of%C2%A0early%C2%A0complementary+feeding%C2%A0on%C2%A0nutritional%C2%A0status+in+term+infants+in+rural+Nigeria.